CLINICAL TRIAL: NCT06593379
Title: Pilot Randomized Controlled Trial of the Mobile Intervention for Suicidal Thoughts
Brief Title: Mobile Intervention for Suicidal Thoughts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5137-P
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Suicide
Keywords: suicide; suicide cognitions; mobile intervention; veterans
MeSH Terms: conditions — Suicide | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 50 Veterans with suicidal ideation will be randomized to either MIST plus Treatment as Usual and Safety Planning versus Treatment as Usual and Safety Planning
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessors will be blinded to the participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safety planning, treatment as usual, and MIST (Experimental): Participants will get a safety plan, treatment as usual, and the MIST intervention.
  Interventions: Behavioral: Safety planning; Behavioral: Treatment as usual; Behavioral: MIST Intervention
- Safety planning and treatment as usual (Active Comparator): Participants will get a safety plan and treatment as usual.
  Interventions: Behavioral: Safety planning; Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Safety planning — Safety planning (SP) is a single-session intervention that consists of developing a written list of individualized coping strategies and sources of support that can be used during a suicidal crisis.
Behavioral: Treatment as usual — This will include continued care with any of the Veterans' current providers. Study staff will also place appropriate referrals for Veterans, as needed (e.g., Trauma Recovery Program referrals for Veterans with PTSD, Sleep Psychology referrals for Veterans with insomnia). Participants will be encouraged to follow up with their providers' recommendations and treatment plans
Behavioral: MIST Intervention — This is a mobile intervention designed to target and modify suicidal cognitions. Veteran in this condition will be asked to use the intervention 5 times a week for 4 weeks.
  Arms: Safety planning, treatment as usual, and MIST

SUMMARY:
One of the factors that contributes to suicide risk is what is known as a "suicidal belief system." This belief system is made up of several cognitions that been associated with suicide risk among military personnel. Modification of these cognitions may reduce suicidal thoughts and behaviors. The study team has developed a brief mobile intervention entitled the Mobile Intervention for Suicidal Thoughts (MIST) that uses evidence-based interpretation bias modification techniques to reduce these suicide cognitions. The goal of this project is to is to conduct a pilot trial of the MIST intervention to evaluate whether it is feasible an acceptable as an adjunct treatment for Veterans with suicidal ideation.

DETAILED DESCRIPTION:
One of the factors that contributes to suicide risk is what is known as a "suicidal belief system." This belief system is made up of several cognitions, including hopelessness, thwarted belongingness, perceived burdensomeness, unlovability, unbearability, and unsolvability. These cognitions have all been associated with suicide risk among military personnel. Modification of these cognitions may reduce suicidal thoughts and behaviors. The study team has developed a brief mobile intervention entitled the Mobile Intervention for Suicidal Thoughts (MIST) that uses evidence-based interpretation bias modification techniques to reduce these suicide cognitions. The goal of this project is to is to conduct a pilot trial of the MIST intervention to evaluate whether it is feasible an acceptable as an adjunct treatment for Veterans with suicidal ideation.

The investigators will conduct a pilot randomized controlled trial (RCT), in which 50 Veterans with suicidal ideation will be randomized to either MIST plus Treatment as Usual and Safety Planning versus Treatment as Usual and Safety Planning. The central hypothesis is that Veterans will find MIST acceptable and will be willing to use it to reduce their suicidal thoughts.

ELIGIBILITY:
Inclusion Criteria:

* Veterans using the Durham VA Health Care System
* Endorsing suicidal ideation without intent in the last 30 days, established via C-SSRS
* Meet at least every 4 months with a mental health provider, established via chart review chart
* Can read at least 6th grade level material, established by their demonstrated ability to read the consent form and answer basic questions about it

Exclusion Criteria:

* Currently in a period of active psychosis or mania, established via the SCID-5
* Currently meeting criteria for a moderate or severe alcohol or substance use disorder, established via the SCID-5
* Endorsing suicidal intent, established via C-SSRS
* Exhibit current prominent suicidal or homicidal ideation requiring immediate intervention
* Have used the MIST intervention before as part of another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | Through study completion (approximately 18 months)
  Participant feasibility goal will be met if recruitment is 75% or greater of recruitment expectation.
Percentage of enrolled participants who complete the study intervention | Post-treatment visit (approximately one month after enrollment)
  Treatment retention feasibility goal will be met if attrition is no more than 25%.
Patient satisfaction for MIST app: Client Satisfaction Questionnaire | Post-treatment visit (approximately one month after enrollment)
  Patient satisfaction will be assessed with item #7 from the Client Satisfaction Questionnaire. This item is scored on a scale of 1 to 4, with one indicating lower satisfaction and 4 indicating greater satisfaction. The patient satisfaction goal will be met if 80% or greater of participants indicate score a 3 or 4 on this item.
MIST intervention utilization | Post-MIST assessment visit (approximately one month after enrollment)
  MIST utilization goal will be met if MIST app utilization rates are greater than 50% of expected use.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten H Dillon, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No